CLINICAL TRIAL: NCT01595230
Title: Randomized Controlled Trial: Internal Hernias After Gastric Bypass Can be Prevented Safely With Primary Closure of All Mesenteric Defects With Clips
Brief Title: Internal Hernias After Gastric Bypass Can be Prevented Safely With Primary Closure of All Mesenteric Defects With Clips
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Region Zealand (Other)
Responsible Party: Principal Investigator, Sara Kristensen, Doctor, Region Zealand
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SJ-284
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Internal Hernias
Keywords: Internal Hernias; Clips; Gastric Bypass; Avoid
MeSH Terms: conditions — Internal Hernia | interventions — Surgical Instruments; Gastric Bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inertervention group_Clips to avoid internal herniation (Experimental): LRYGB with closure of the defects with simple hernia stapler clips. Aim of this study is to evaluate the benefits and disadvantages of closing the mesenteric defects during gastric bypass in order to avoid internal herniation.
  Interventions: Procedure: Closing the mesenteric defects with clips during opration
- Control group (No Intervention): conventional LRYGB without closure of the mesenteric defects

INTERVENTIONS:
Procedure: Closing the mesenteric defects with clips during opration — The laparoscopic Roux-en-Y gastric bypass surgery will be performed as usual. The patient will receive the closing of the mesenteric defects (the Petersen´s space and the entero-enterostomy site).The closing will happen at the end of the operation, using clips (herniestapler).
  Other Names: Clips, Herniestapler, Internal hernia, Gastric bypass
  Arms: Inertervention group_Clips to avoid internal herniation

SUMMARY:
The purpose of this study is to determine whether closure of all mesenteric defects with clips at the time of Gastric bypass, can avoid the complication of late bowel obstruction- internal hernias

ELIGIBILITY:
Inclusion Criteria:

* All patients who meet the requirements for a Gastric Bypass at Køge Hospital.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria
* Patients who converted to open surgeon

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2012-05; Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
To avoid the risk of Internal Hernias in patient with a Gastric bypass | 5 year

SECONDARY OUTCOMES:
Postoperative pain score (VAS) | 5 years
Operative time consumption, the amount of clips, trocar and sutures used | 3 years

OTHER OUTCOMES:
30 days complication | 3 years
  30 days complications:
  * Anastomotic leak
  * Bleeding (Hb)
  * Blood transfusions (MAF)
  * Ileus due to kinking, blowout of the bypassed stomach
  * Intraperitoneal abscesses.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Kristensen, Doctor, Principal Investigator — Department of Surgery, Bariatric Clinic, Koge Hospital
Locations (2):
- Denmark (2):
  - Department of Surgery;Bariatric Clinic, Køge Hospital, Køge, Sealand
  - Bariatric clinic, Department of Surgery, Køge hospital, Køge

REFERENCES:
- [Derived] Kristensen SD, Gormsen J, Naver L, Helgstrand F, Floyd AK. Randomized clinical trial on closure versus non-closure of mesenteric defects during laparoscopic gastric bypass surgery. Br J Surg. 2021 Mar 12;108(2):145-151. doi: 10.1093/bjs/znaa055. PMID 33711136
- [Derived] Kristensen SD, Naver L, Jess P, Floyd AK. Effect of closure of the mesenteric defect during laparoscopic gastric bypass and prevention of internal hernia. Dan Med J. 2014 Jun;61(6):A4854. PMID 24947625